CLINICAL TRIAL: NCT06728020
Title: ROOMMATE - AggRegated System Of sensOrs and Multimedia Monitors: Technology for innovAtion and personalizaTion of rEhabilitation Care.
Brief Title: AggRegated System Of sensOrs and Multimedia Monitors: Technology for innovAtion and personalizaTion of rEhabilitation Care. (ROOMMATE)
Acronym: ROOMMATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francesca Cecchi (Other)
Collaborators: MEDEA, Italy (Unknown); Carol Davila University of Medicine and Pharmacy (Other); Roessingh Research and Development (Other); University of Florence (Other)
Responsible Party: Sponsor-Investigator, Francesca Cecchi, Associate Professor, Fondazione Don Carlo Gnocchi Onlus
Organization: Fondazione Don Carlo Gnocchi Onlus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: cmRCT ROOMMATE; Grant Agreement Nº: 101095654. (Other Grant/Funding Number: Tranforming Health and Care Systems partnership)
Record Dates: First submitted 2024-11-27; First posted 2024-12-11 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Subacute Stroke; Stroke; Subacute
Keywords: subacute stroke; Neurorehabilitation; Assistive/rehabilitation robotics; Digital health; Continuum of care; People-centered care; Accessible care; Innovation adoption; cmRCT; Enriched environment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Three phases: in the first, focus groups and living labs are conducted to co-create the solution with patients; in the second, as the first action of the cmRCT, an RCT is conducted to verify the effectiveness of the initial ROOMMATE system; in the third, a pilot is conducted to preliminarily test the advanced version of the ROOMMATE system.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional rehabilitation (Group A) (Active Comparator): The first 140 patients who meet the inclusion criteria will be randomized between this group and group B. This group will undergo conventional therapy.
  Interventions: Other: Active Comparator: Conventional rehabilitation (Group A)
- ROOMMATE 1st (Group B) (Experimental): The 70 patients randomized to this group will undergo conventional treatment and, in addition, will have the first version of the ROOMMATE system.
  Interventions: Device: ROOMMATE 1st
- ROOMMATE 2nd (Goup B2) (Experimental): Group B2 will undergo conventional treatment and will have an extended version of the bedside multimedia monitor apparatus, integrated with an inertial sensor to enable the serious games on the experimental platform.
  Interventions: Device: ROOMMATE 2nd

INTERVENTIONS:
Other: Active Comparator: Conventional rehabilitation (Group A) — The conventional group will undergo standard rehabilitation treatment according to the rehabilitation plan developed by the rehabilitation team. This group will undergo 3 hours of rehabilitation per day and will carry out face-to-face rehabilitation following an impairment-based approach aimed at the treatment of motor-cognitive functions.
  Arms: Conventional rehabilitation (Group A)
Device: ROOMMATE 1st — In addition to Group A, this group will have the bedside multimedia monitor apparatus to access informative, rehabilitation, and entertainment content. Additionally, this group will have a digital and innovation coach to receive support in using the technology.
  Arms: ROOMMATE 1st (Group B)
Device: ROOMMATE 2nd — Once the first RCT of the cmRCT is completed, a pilot RCT will be initiated, randomizing 60 cases between Group A and this group. In addition to conventional treatment, this group will have a version of the ROOMMATE system integrated with inertial sensors worn on the hands and fingers to guide the serious games on the platform.
  Arms: ROOMMATE 2nd (Goup B2)

SUMMARY:
The aim of this clinical trial is to assess whether the ROOMMATE system can effectively support the rehabilitation of adults recovering from subacute strokes. The study will be conducted at the neuromotor rehabilitation inpatient clinics of IRCCS Fondazione Don Carlo Gnocchi in Florence, Italy, and the rehabilitation inpatient unit of Elias University Emergency Hospital in Bucharest, Romania.

Primary Objectives:

-To assess the effects on functional recovery in subacute stroke survivors of a technological rehabilitation station placed at patients' bedsides, combined with dedicated coaching provided to all users (patients, informal caregivers, and formal caregivers).

Secondary Objectives:

* Evaluation of the effects of the experimental treatment on patient satisfaction, upper limb motor skills, manual dexterity, global cognitive functioning, anxiety, and depression.
* Assessment of user experience, acceptance, and usability of the technology by patients and caregivers.
* Evaluation of social impact using the Social Return on Investment (SROI) ratio of the experimental treatment.

Participants randomized into one of the experimental groups, in addition to receiving conventional care, will use the ROOMMATE system during their hospitalization. The system will be made available to patients and will be free for them to use at their discretion.

The station will include:

Multimedia monitors (Khymeia home kit): These will deliver cognitive and motor serious games, educational and rehabilitative content, as well as infotainment specifically developed by the clinical partners of the project.

An inertial sensor kit: This integrates with the monitors to guide users through virtual reality environments.

DETAILED DESCRIPTION:
Study Procedures

The study involves three successive phases:

Phase 1 During the first phase, after obtaining Ethics Committee approval, Living Labs will be planned. In these sessions, end users will test the proposed solutions and provide feedback on acceptability and usability. This phase is critical for defining user and system requirements. Additionally, health professionals will be trained as system coaches to support patients and their families in the subsequent phases.

The coaches will be selected from health professionals (physical therapists, occupational therapists, speech therapists, psychologists, nurses) with at least three professionals per center. They will complete a one-week course in digital literacy (e-literacy), covering:

* Technical and operational skills for managing and using digital technologies.
* Information and navigation skills.
* Specific training on the use of the Khymeia Home Kit.
* Training on using the inertial sensors developed by UNIFI. The training will conclude with a written and practical exam.

Subsequently, a multicenter multiple cohort RCT (cmRCT) will be conducted, consisting of two trials:

1. A first RCT (Phase 2 of the study).
2. A second pilot RCT (Phase 3 of the study). The study will be carried out in an inpatient setting for individuals with subacute stroke outcomes at the two clinical centers: IRCCS Fondazione Don Carlo Gnocchi in Florence, Italy, and Elias University Emergency Hospital in Bucharest, Romania.

The cmRCT design was chosen to address some limitations of traditional RCTs, such as issues with recruitment, ethics, patient preferences, and treatment comparison. Moreover, the cmRCT allows the simultaneous evaluation of different interventions.

In ROOMMATE, eligible patients who consent to baseline (T0) and final (T1, three weeks later) assessments may also be offered an additional intervention, forming the ROOMMATE Study Cohort. A subset of these patients will be randomized to receive an offer to participate in the ROOMMATE Interventions (B or B1), while those not randomized will form the control group (A, receiving usual care). This design will allow two successive RCTs to be conducted.

Phase 2

The first RCT will compare usual care (A) with a preliminary version of the ROOMMATE solution (B), which includes:

* Usual care.
* The Khymeia Home Kit monitor.
* Educational and rehabilitative content developed by clinical partners.
* Coaching for technology use. The sample size for this RCT is 140 patients, randomly assigned to Group A or B, with competitive enrollment across the two clinical centers.

The Khymeia Home Kit, supplemented with educational content, can be used by patients alone or with a caregiver. The educational materials will include:

* General information about stroke pathogenesis and prognosis.
* Strategies and advice for managing the condition.
* Health-related content, such as details on daily hospitalization routines, the roles of various care professionals, and discharge management (including bureaucratic aspects).
* Information on local support networks. Additional cognitive and motor rehabilitation content will be developed by a multidisciplinary team and customized by department therapists to match each patient's needs and recovery potential.

The coach will be available in person five days a week to support all end users in using the ROOMMATE technology.

Phase 3

Following the completion of the first RCT, a second pilot RCT with 60 patients will test usual care (A) against a mature version of the ROOMMATE solution (B1). This includes:

* Usual care.
* Motor and cognitive treatment supported by inertial sensor assessment for personalized interventions.
* Integration of clinical assessments with IMU-derived reports.
* Educational and rehabilitative content developed by clinical partners.
* Coaching for technology use. In Group B1, the Khymeia Home Kit (with educational and rehabilitation content) will be enhanced with inertial sensors developed by UNIFI. These sensors will measure hand motility and provide tailored rehabilitation interventions.

The ROOMMATE intervention will last three weeks per patient. During this period:

* Group B patients will receive training in using the technology from the coach.
* Patients and their families will have self-directed or supervised access to HKK features, including educational, rehabilitative, and infotainment content.
* Therapists will recommend the most appropriate content based on the patient's needs.
* In Group B1, the physician will use inertial sensor data to quantify motor deficits and tailor the treatment accordingly.

Assessments (T0 and T1)

At baseline (T0) and post-treatment (T1), the following will be assessed:

* Demographics: Sex, age, education.
* Clinical data: Type of stroke, time since stroke, lesion laterality.
* Primary and secondary outcomes: Disability in ADLs (modified Barthel Index, mBI). Manual dexterity. Upper limb motor skills. Neuropsychological and global cognitive functioning. Anxiety and depression. Quality of life.

At post-treatment (T1), also the following will be assessed:

• Primary and secondary outcomes: Usability, feasibility, and social impact measures. User experience and education evaluation. Wearability of sensors. Social impact and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* outcome of ischemic or hemorrhagic stroke in subacute phase (< 3 months after the event)
* willingness to participate in the project, with informed consent signed by the subject or, when necessary, by the support administrator.

Exclusion Criteria:

* severe visual and/or auditory impairments that cannot be corrected
* severe cognitive and/or speech impairments that interfere with the ability to use the HKK system and the SensoMode accessory independently and/or in the
* absence of a caregiver who can assist the patient in using the system;
* skin lesions that prevent wearing the inertial sensors;
* presence of signs of clinical instability, defined by a score greater than zero on the Clinical Instability Scale (SIC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
modified Barthel index (mBI) | baseline, 3 week
  Assessment of disability in ADLs, scoring 0-100

SECONDARY OUTCOMES:
Nine Hole Peg Test | baseline, 3 week
  Manual Dexterity, evaluated in seconds
Fugl Meyer Assessment (FMA) | baseline, 3 week
  Upper limb motor skills, scoring 0 - 126
Functional Ambulation Category (FAC) | baseline, 3 week
  functional ambulation assessment, scoring 0-5
Montreal Cognitive Assessment (MOCA) | baseline, 3 week
  Cognitive impairment assessment, scoring 0 - 30
Hearts Test | baseline, 3 week
  3-minute visual attention barrage test, scores 0-50
Short Form 12 item | baseline, 3 week
  generic assessment of quality of life, scoring 0-47
Training-Evaluation-Inventory (TEI) | 3 week
  evaluation of the course and its contents, a 45 item scale scoring with a 5 point likert scale
Short Version of the User Experience Questionnaire (UEQ-S) | 3 week
  user expirience assessment, 8 item scale scoring with a 7 point likert scale
Final Measurement Scales for Perceived Usefulness and Perceived Ease of Use | 3 week
  Acceptance Assessment of the ROOMATE sistem, a 12 item scale scoring with a 7 point likert scale
HUBBI - eHealth UsaBility Benchmarking Instrument | 3 week
  Usability Assessment of the ROOMATE sistem, a 18 item scale scoring with a 5 point likert scale
we wearability test | 3 week
  Sensors Wearability Assessment, likert scale, scores 1-5
Motricity Index | baseline, 3 week
  Upper limb and lower limb motor skills, scoring 0 - 100

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi Onlus, Florence, Florence, Italy

IPD SHARING:
Plan to Share IPD: Yes
After publishing the results in international congresses and conferences and in impacted journals, the project partners, according to the stipulated data management plan will disseminate the results following the principle of "as open as possible, as closed as needed". Resuls will be shared on a Zenodo-like repository.
Supporting Information: Study Protocol, CSR
Time Frame: We plan to share:
  * preliminary results as the study progresses.
  * The study protocol on an international impacted journal upon obtaining ethics committee and the number of registration on clinicaltrials.gov.
  * The study results, within two year, at the end of the study

REFERENCES:
- [Derived] Doronzio S, Jansen-Kosterink S, Tesi M, Castagnoli C, Pedrini C, Ciapetti T, De Marco M, Piazzini M, Giacani J, Ciobanu I, Berteanu M, Fiorini L, Rovini E, Cavallo F, Agnoloni F, Baccini M, Cecchi F. Development of a cohort multiple randomized clinical trial to test an integrated system of sensors and multimedia monitors technology, for stroke rehabilitation: the ROOMMATE study protocol. Front Neurol. 2025 Oct 14;16:1568728. doi: 10.3389/fneur.2025.1568728. eCollection 2025. PMID 41164394